CLINICAL TRIAL: NCT01238913
Title: Prospective Evaluation of the Clinical Utility of the Endoscopic Placement of Mental Stent for Benign Esophageal Lesions
Brief Title: Use of Metal Stents on Benign Esophageal Lesions
Status: Withdrawn | Type: Observational
Why Stopped: No one met the inclusion/exclusion criteria
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Benign esophageal lesions
Record Dates: First submitted 2010-11-05; First posted 2010-11-11 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Benign Esophageal Lesions
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- benign esophageal lesions: All patients who have a benign esophageal lesion where it is medically indicated that they receive a stent.
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Endoscopic placement of an esophageal metal stent as per medical indication.

SUMMARY:
The evaluation of using metal stents as medically indicated for the treatment of benign esophageal lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject has medical indication to undergo endoscopic placement of esophageal metal stent
3. Subject must be able to give informed consent

Exclusion Criteria:

1. Any contraindications for endoscopic placement of esophageal metal stent
2. The subject is unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a medical indication for endoscopic placement of esophageal metal stent and are referred for the porcedure as part of their standard medical care will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Successful stenting of Benign esophageal lesions | approximately 2-3 hours
  This is an observational study to determine the effectiveness of stenting benign esophageal lesions with a metal stent.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida